CLINICAL TRIAL: NCT06845683
Title: Effects of Dual-Task and Progressive Wall Squat Training on Cognition, Balance and Functional Mobility in Stroke Survivors
Brief Title: Effects of Dual-Task and Progressive Wall Squat Training in Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/24/0211 Barira Shahid
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Stroke Ischemic
Keywords: Balance; cognition; dual-task; functional mobility; stroke survivors; wall squat
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and outcome assesssors wtll be kept blinded about the intervention which the patients will be going to receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combining progressive wall squats with cognitive training (Experimental): Group A will receive dual-task intervention (combining progressive wall squats with cognitive training) along with routine rehabilitation. The group will undergo 45 minute treatment session three times per week over an eight weeks period, focusing on gradually intensifying the progressive wall squat exercises with careful supervision to ensure safety and proper form along with cognitive tasks.
  Interventions: Other: Group A
- progressive wall squats (Active Comparator): Group B will receive single-task intervention (involving progressive wall squats) along with routine rehabilitation. A routine rehabilitation comprising slow sustained stretching (with a hold time of 10 seconds per stretch, totaling 10 repetitions per session) and active range of motion exercises (10 repetitions per session) targeting both the upper and lower extremities. The group will undergo 45 minute treatment session three times per week over an eight weeks period.
  Interventions: Other: Group B

INTERVENTIONS:
Other: Group A — Progressive wall squat exercises will commence with a knee flexion angle of 135°, instructed to hold this position for 20 seconds, exercise progresses, the knee joint angle will be decreased by 10° until reaching the 95° stage or until participants can no longer maintain the knee joint angle within 5° of the target value due to volitional fatigue. Cognitive tasks during the intervention, including the recall of words and counting forward (1, 4, 7, 10...) and backward (...10, 7, 4, 1) by adding 3 to the digits. Sustained stretching (with a hold time of 10 seconds per stretch, totaling 10 repetitions per session) and active range of motion exercises (10 repetitions per session) targeting both the upper and lower extremities in routine rehabilitation.
  Other Names: Dual task training (Wall squats + cognitive training along with routine rehabilitation
  Arms: combining progressive wall squats with cognitive training
Other: Group B — Progressive wall squat exercises will commence with a knee flexion angle of 135°, instructed to hold this position for 20 seconds, exercise progresses, the knee joint angle will be decreased by 10° until reaching the 95° stage or until participants can no longer maintain the knee joint angle within 5° of the target value due to volitional fatigue. Sustained stretching (with a hold time of 10 seconds per stretch, totaling 10 repetitions per session) and active range of motion exercises (10 repetitions per session) targeting both the upper and lower extremities in routine rehabilitation.
  Other Names: single-task intervention (Wall squats) along with routine rehabilitation
  Arms: progressive wall squats

SUMMARY:
To determine the Effects of Dual-Task and Progressive Wall Squat Training on Cognition, Balance and Functional mobility in Stroke Survivors.

DETAILED DESCRIPTION:
A stroke is a neurological disorder in which clots or ruptured vessels obstruct blood vessels, causing abnormal blood flow in the brain. This may lead to the unexpected death of brain cells and aggravate illnesses like depression and dementia.It is a disease with significant health and social consequences because of its high frequency and rate. Stroke is thought to affect 9.2% of the population in Europe, with a rate of 191.9 per 100,000 people annually. According to estimates, between 25 and 74% of those who survive this illness need assistance or become totally reliant on their everyday activities.The primary long-term effects of a stroke are dysphagia, paralysis, motor impairments, cognitive decline, and speech difficulties.

Dual-task training entails doing a motor task and a cognitive task at the same time. This method's justification is that a lot of daily tasks necessitate multitasking, and dual-task training can improve both cognitive and motor abilities by promoting brain plasticity and the interaction of the two systems. In the dual task training, cognitive task (like naming animals or counting backwards) is combined with a lower limb strengthening exercise called wall squats. Both tasks gradually increase in difficulty and intensity based on how well each person performs. By testing the muscle strength, endurance, and coordination of stroke survivors as well as their attention, memory, and executive function, this training seeks to improve their cognitive abilities, balance, and functional mobility.

ELIGIBILITY:
Inclusion Criteria:

* Age: Stroke patients aged 45 to 65 years.
* Individuals with a single ischemic stroke.
* Within the first 2 months post-stroke. (Subacute stage)
* Medically stable without acute conditions interfering with exercise.
* Mini-Mental State Examination (MMSE) score≥24
* Ability to walk 10m without assistance

Exclusion Criteria:

* Unstable Medical Conditions (cardiovascular, respiratory, or other medical conditions)
* Recent Stroke or Medical Event
* Other Neurological Conditions such as Presence of other neurological conditions (e.g., Parkinson's disease).
* Uncontrolled Hypertension: Systolic BP >160 mm Hg or diastolic BP >100 mm Hg

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
MOCA (Montreal Cognitive Assessment) | 8 weeks
  A well-liked screening method for identifying the presence of cognitive impairment is the MoCA. It takes about ten minutes to finish. It assesses language, abstract reasoning, executive function, orientation, delayed recall, attention, and visuospatial skills. The MoCA is more sensitive and specific than the MMSE because it covers a wider range of domains.
Tinneti POMA (Balance, gait) | 8 weeks
  The Tinetti Scale is a tool for assessing gait and balance. The test is used clinically to evaluate changes in gait time and balance, as well as to ascertain a subject's current level of mobility. The two sub-scales that make up the total POMA (POMA-T) are the gait evaluation scale (also known as the POMA-G) and the balance evaluation scale (also known as the POMA-B). The maximum score is 28 points; specifically, the POMA-B has a maximum score of 16 and the POMA-G has a maximum score of 12.
Rivermead mobility index | 8 weeks
  RMI is a measure that evaluates a patient's degree of mobility .There are 14 questions on it, along with a section on observations. This index evaluates an individual's ability to do tasks like getting out of bed, sitting, maintaining balance, standing up, standing unassisted, moving around, walking indoors and outside, climbing and descending stairs, picking up objects off the floor, taking a shower, and running. Every activity receives one point, if at all possible. If the score is less than 14, it suggests that the person has mobility problems; if the score is 15, it means they don't have any problems at all

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Riphah International University Pakistan
Locations (1):
- Society Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morice E, Moncharmont J, Jenny C, Bruyneel AV. Dancing to improve balance control, cognitive-motor functions and quality of life after stroke: a study protocol for a randomised controlled trial. BMJ Open. 2020 Sep 30;10(9):e037039. doi: 10.1136/bmjopen-2020-037039. PMID 32998921
- [Background] Buvarp D, Rafsten L, Sunnerhagen KS. Predicting Longitudinal Progression in Functional Mobility After Stroke: A Prospective Cohort Study. Stroke. 2020 Jul;51(7):2179-2187. doi: 10.1161/STROKEAHA.120.029913. Epub 2020 Jun 17. PMID 32568652
- [Background] Lee Y, Kim K. The influence of Gait Training Combined with Portable Functional Electrical Stimulation on motor function, balance and gait ability in stroke patients. J Back Musculoskelet Rehabil. 2022;35(6):1171-1178. doi: 10.3233/BMR-210154. PMID 35754258
- [Background] Hurd MD, Goel I, Sakai Y, Teramura Y. Current status of ischemic stroke treatment: From thrombolysis to potential regenerative medicine. Regen Ther. 2021 Oct 12;18:408-417. doi: 10.1016/j.reth.2021.09.009. eCollection 2021 Dec. PMID 34722837
- [Background] Spano B, Lombardi MG, De Tollis M, Szczepanska MA, Ricci C, Manzo A, Giuli S, Polidori L, Griffini IA, Adriano F, Caltagirone C, Annicchiarico R. Correction: Spano et al. Effect of Dual-Task Motor-Cognitive Training in Preventing Falls in Vulnerable Elderly Cerebrovascular Patients: A Pilot Study. Brain Sci. 2022, 12, 168. Brain Sci. 2024 Apr 11;14(4):370. doi: 10.3390/brainsci14040370. PMID 38672060
- [Background] Kuriakose D, Xiao Z. Pathophysiology and Treatment of Stroke: Present Status and Future Perspectives. Int J Mol Sci. 2020 Oct 15;21(20):7609. doi: 10.3390/ijms21207609. PMID 33076218